CLINICAL TRIAL: NCT04471415
Title: Phase 1 and Phase 2a, First-in-human Study of DRP-104, a Glutamine Antagonist, in Adult Patients With Advanced Solid Tumors
Brief Title: Study to Investigate DRP-104 in Adults With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company decision to closing study and discontinue further patient enrollment.
Sponsor: Dracen Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DRA-104-001; 2020-002770-27 (EudraCT Number)
Record Dates: First submitted 2020-06-25; First posted 2020-07-15 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Advanced Solid Tumor; Non Small Cell Lung Cancer Metastatic
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: Dose Escalation cohort, followed by Dose Expansion cohort, followed by NSCLC, and in combination with atezolizumab cohorts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1a & Part 1b (Experimental): Single-agent dose escalation of DRP-104 to define the MTD (up to approximately 50 patients) starting at Dose Level 1 of 3.3 mg/m2 via intravenous injection
  Single-agent dose escalation of DRP-104 to define the MTD (up to approximately 50 patients) starting at Dose Level 1 at 10 mg via subcutaneous injection
  Interventions: Drug: DRP-104
- Part 2 (Experimental): Cohort 1: Phase 1 single-agent safety expansion of DRP-104 administered subQ (the RP2R) in patients with advanced solid tumors (excluding primary CNS tumors and HCC). DRP-104 will be administered twice weekly subQ in this safety expansion at the twice weekly subQ MTD/MAD/RP2D of DRP-104 determined in Part 1-Cohort 1b. A minimum of 14 and up to 20 patients will be enrolled.
  Cohort 2: Phase 2a expansion at the MTD/MAD/RP2D/RP2R and schedule of administration (subQ twice or thrice weekly) of DRP-104 in patients with locally advanced or metastatic NSCLC whose tumors contain a known mutation in kelchlike ECH-associated protein 1 (KEAP1), nuclear factor erythroid 2-related factor 2 (NFE2L2) and/or serine/threonine kinase 11 (STK11), (N=55). If the thrice weekly schedule is selected as the RP2S, a safety review will be conducted after 8 patients have enrolled and are followed for at least one cycle of treatment before additional patients are enrolled into Part 2-Cohort 2.
  Interventions: Drug: DRP-104
- Part 3 (Experimental): Phase 1 combination dose escalation of DRP-104 and atezolizumab in patients with advanced solid tumors (excluding primary CNS tumors and HCC) previously treated with an agent targeting checkpoint pathway inhibition (such as anti-PD-1, anti-PD-L1, and/or anti-CTLA-4 antibody), starting one dose level below the MTD/MAD/RP2D (MTD-1) of the recommended phase 2 route and schedule of administration of singleagent DRP-104 and in combination with 1200 mg atezolizumab administered via intravenous infusion on day 1 and repeated every 3 weeks (up to approximately 12 patients);
  Interventions: Drug: DRP-104; Biological: atezolizumab
- Part 4 (Experimental): Phase 1 combination safety expansion at the MTD/MAD/RP2D, route, and schedule of administration of DRP-104 with atezolizumab in a similar patient population as the dose-escalation (N=14 patients).
  Interventions: Drug: DRP-104; Biological: atezolizumab

INTERVENTIONS:
Drug: DRP-104 — DRP-104 administered intravenously over 1 hour, three times per week (TIW) (Monday, Wednesday, Friday) for 2 consecutive weeks, one week off
  DRP-104 administered subcutaneously twice weekly (Monday/Thursday or Tuesday/Friday) every week OR thrice weekly (Monday, Wednesday, Friday) every week
Biological: atezolizumab — atezolizumab administered intravenously over 1 hour at 1200 mg once every 3 weeks.
  Arms: Part 3; Part 4

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, pharmacokinetics, pharmaco-dynamics and preliminary anti-tumor activity of DRP-104 (sirpiglenastat) administered via intravenous infusion or via subcutaneous injection as a single agent and in combination with atezolizumab in patients with advanced solid tumors and to assess preliminary safety and efficacy of which route of administration (intravenous or subcutaneous) will be selected for further development for the one expansion of patients, advanced non-small cell lung cancer (NSCLC) with defined genetic mutations.

DETAILED DESCRIPTION:
This study will be conducted in 4 Parts:

Part 1: Phase 1 single-agent dose escalation of DRP-104 administered via IV infusion (Cohort 1a) or subQ injection (Cohort 1b and 1c) in patients with advanced solid tumors (excluding primary CNS tumors and HCC):

1. Cohort 1a: IV DRP-104 dose escalation to define the IV MTD/MAD/RP2D (up to approximately 50 patients)
2. Cohort 1b: subQ twice weekly DRP-104 dose escalation to define the twice weekly subQ MTD/MAD/RP2D (up to approximately 50 patients)
3. Cohort 1c: subQ thrice weekly DRP-104 dose escalation to define the thrice weekly subQ MTD/MAD/RP2D (up to approximately 12 patients) Upon completion of Part 1, Cohort 1a, 1b, and 1c, the recommended phase 2 route of administration (RP2R: IV or subQ) and schedule of administration (RP2S: twice or thrice weekly) and corresponding MTD/MAD/RP2D will be determined prior to starting Part 2, cohort 2. As of Version 5 of the protocol, further assessment of the intravenous formulation was terminated prior to declaring MTD/MAD/RP2D and the RP2R was determined to be subQ (Section 2.5.5).

Part 2, which opens to enrollment once the MTD/MAD/RP2D/RP2R of DRP-104 has been declared from either Part 1-Cohort 1a, 1b, or 1c and/or the RP2R/RP2S has been determined from Part 1 and includes 2 specific cohorts:

1. Cohort 1: Phase 1 single-agent safety expansion of DRP-104 administered subQ (the RP2R) in patients with advanced solid tumors (excluding primary CNS tumors and HCC). DRP-104 will be administered twice weekly subQ in this safety expansion at the twice weekly subQ MTD/MAD/RP2D of DRP-104 determined in Part 1-Cohort 1b. A minimum of 14 and up to 20 patients will be enrolled.
2. Cohort 2: Phase 2a expansion at the MTD/MAD/RP2D/RP2R and schedule of administration (subQ twice or thrice weekly) of DRP-104 in patients with locally advanced or metastatic NSCLC whose tumors contain a known mutation in kelchlike ECH-associated protein 1 (KEAP1), nuclear factor erythroid 2-related factor 2 (NFE2L2) and/or serine/threonine kinase 11 (STK11), (N=55). If the thrice weekly schedule is selected as the RP2S, a safety review will be conducted after 8 patients have enrolled and are followed for at least one cycle of treatment before additional patients are enrolled into Part 2-Cohort 2.

Part 3: Phase 1 combination dose escalation of DRP-104 and atezolizumab in patients with advanced solid tumors (excluding primary CNS tumors and HCC) previously treated with an agent targeting checkpoint pathway inhibition (such as anti-PD-1, anti-PD-L1, and/or anti-CTLA-4 antibody), starting one dose level below the MTD/MAD/RP2D (MTD-1) of the recommended phase 2 route and schedule of administration of singleagent DRP-104 and in combination with 1200 mg atezolizumab administered via intravenous infusion on day 1 and repeated every 3 weeks (up to approximately 12 patients); The dose of atezolizumab is fixed. Enrollment for Part 3 will begin once at least 14 patients from either Part 1 or 2 have been treated at this dose, route, and schedule for at least one cycle to ensure safety.

Part 4: Phase 1 combination safety expansion at the MTD/MAD/RP2D, route, and schedule of administration of DRP-104 with atezolizumab in a similar patient population as the dose-escalation (N=14 patients).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced or recurrent, histologically or cytologically confirmed, measurable by RECIST 1.1 metastatic or unresectable solid tumor
* Patient must have progressed on, be intolerant of, decline, or be ineligible for, all available standard of care therapies
* Part 2: locally advanced or metastatic NSCLC with KEAP1, NFE2L2 and/or STK11 mutation ; Patients must have received at least a platinum doublet chemotherapy and an anti-PD-(L)1 antibody; Received up to 3 lines of systemic anticancer therapy in the recurrent or metastatic setting
* Part 3 and 4 - DRP-104 + atezolizumab Prior exposure to any checkpoint inhibitor (anti-PD-1, anti-PD-L1, anti-PDL2, and/or anti-CTLA-4 antibody)
* ECOG performance 0 or 1
* Patient must consent to allow acquisition of existing FFPE tumor tissue; If unavailable, patient must consent to new pre-treatment tumor biopsy
* All SCCHN patient, all NSCLC patients and all patients treated with combination of DRP-104 and atezolizumab will be required to undergo pre-treatment and post-treatment core or excisional biopsies.
* Pre-treatment and post-treatment core or excisional biopsies are optional for all remaining patients
* Adequate baseline organ function as defined by: Absolute neutrophil count ≥ 1.5 × 109/L (1500/µL); Hemoglobin ≥ 9 g/dL (patients that require transfusion or growth factors need to demonstrate stable hemoglobin of ≥ 9 g/dL over at least a 7-day period after the last transfusion/growth factor injection prior to screening labs to meet eligibility) ; Platelets ≥ 75 × 109/L (75,000/µL); Hepatic Total bilirubin ≤1.5 × upper limit of normal (ULN): PT/INR and PTT ≤1.5 × ULN, unless treated with warfarin; AST(SGOT)/ALT(SGPT) ≤3 × ULN or ≤ 5 × ULN for patients with liver metastases; Creatinine clearance ≥ 60 ml/min/1.73m2 measured or calculated
* Cardiac QTc (Fridericia) <470 ms
* Women of child-bearing potential and men who are sexually active must agree to use one highly effective method of contraception

Exclusion Criteria:

* Patients with primary central nervous system tumors and hepatocellular carcinoma
* Patients with progressive or symptomatic brain metastases or leptomeningeal disease
* Patients who have not recovered to grade 1 or baseline from adverse events (CTCAE v 5.0) related to prior therapy excluding alopecia, peripheral neuropathy and ototoxicity, which are excluded if ≥ grade 3.
* Lymphopenia ≤ grade 3 is allowed if not related to prior anticancer therapy. If related to prior anticancer therapy, lymphopenia must resolve to ≤ grade 1 or baseline.
* Spinal cord compression not definitively treated with surgery and/or radiation
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage
* Prior glutaminase inhibitor use
* Prior systemic anticancer treatment (i.e., chemotherapy, biologic therapy, monoclonal antibodies, investigational agents) within 21 days or 5 half-lives, whichever is shorter
* Anti-androgen therapies for prostate cancer, such as bicalutamide, within 4 weeks prior to enrollment
* Patients must have recovered from all AEs due to previous therapies to CTCAE v 5.0 grade 1 or baseline, excluding, alopecia, peripheral neuropathy and ototoxicity, which must be at least grade 2 or baseline
* Prior small port palliative radiotherapy within 14 days of start of Cycle 1
* Any major surgery within 21 days from start of Cycle 1
* Secondary malignancy that is progressing or has required active treatment within the past 3 years, except basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy
* Has a known history of HIV or HBV
* Gastrointestinal (GI) function impairment or GI disease
* Significant, uncontrolled heart disease and/or cardiac repolarization abnormality
* Exclusion specific to only Part 3 and 4 (DRP-104 combined with atezolizumab):
* History of severe allergic, anaphylactic to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells
* Prior anti-PD-1, anti-PD-L1 and/or anti CTLA4- agent, patient must not have had a serious (> Grade 3) immune-related AE requiring treatment
* History of autoimmune disease except hypothyroidism on thyroid replacement hormone therapy, idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis
* Patients with underlying condition requiring systemic corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications or other systemic immunosuppressant medications may be enrolled in the study after approval by the Medical Monitor
* History of organ transplantation and/or hematopoietic stem cell transplantation
* Evidence or history of active or latent tuberculosis infection
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1 Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | anticipated 2 year
  Safety
Pharmacokinetics (PK) of DRP-104 | anticipated 1 year
  To assess and compare the concentration and partitioning of DRP-104 and the metabolites M1 and DON
Cmax of DRP-104 | anticipated 1 year
  Area under the plasma concentration versus time curve (AUC)
Overall Response Rate (ORR) | anticipated 2 years
  Using RECIST criteria, determine the Overall Response Rate for DRP-104 subQ in NSCLC cohort 2 (months)

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | anticipated 2 years
  Disease Control Rate of all patient cohorts (months) for IV and SubQ administration
Progression-Free Survival (PFS) | anticipated 2 years
  Using RECIST criteria to assess the time for the disease to progress during treatment with DRP-104 (months)
Overall Survival (OS) | anticipated 2 years
  Defined as the time (months) from the start of treatment to death

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Sharma, MD, Principal Investigator — HonorHealth Director
Locations (22):
- United States (13):
  - HonorHealth, Scottsdale, Arizona
  - UCLA, Los Angeles, California
  - AdventHealth Medical Group, Kissimmee, Florida
  - Florida Cancer Specialist, Orlando, Florida
  - Johns Hopkins Kimmel Institute, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - NYU Langone, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - NEXT Oncology, Fairfax, Virginia
- Germany (4):
  - Centrum fur Integrieerte Onkologie, Cologne
  - University Cancer Center NCT, Dresden
  - University Hospital Frankfurt, Frankfurt
  - University Klinikum Wuerzburg, Würzburg
- National Cancer Center Singapore, Singapore, Singapore
- Spain (2):
  - Hospital University Vall d'Hebron, Barcelona
  - University Hospital 12 de Octubre, Madrid
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Encarnacion-Rosado J, Sohn ASW, Biancur DE, Lin EY, Osorio-Vasquez V, Rodrick T, Gonzalez-Baerga D, Zhao E, Yokoyama Y, Simeone DM, Jones DR, Parker SJ, Wild R, Kimmelman AC. Targeting pancreatic cancer metabolic dependencies through glutamine antagonism. Nat Cancer. 2024 Jan;5(1):85-99. doi: 10.1038/s43018-023-00647-3. Epub 2023 Oct 9. PMID 37814010
- See also: Company website with scientific background on DRP-104 — http://www.dracenpharma.com/